CLINICAL TRIAL: NCT01164761
Title: A Two-way Open Label Crossover Experimental Evaluation of Relative Bioavailabilities of Ramipril 10 mg Capsules of Dr.Reddy's Laboratories and ALTACE@ 10 mg Capsules of King Pharmaceuticals in Healthy Adult Human Male Subjects Under Fasting Conditions
Brief Title: Bioavailability Study of Ramipril 10 mg Capsules of Dr. Reddy's Laboratories Limited Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Mr. M.S. Mohan / Senior Manager R & D, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 074-05
Record Dates: First submitted 2010-07-16; First posted 2010-07-19 (Estimated); Last update posted 2010-07-19 (Estimated); Status verified 2010-07

CONDITIONS: Healthy
Keywords: Bioavailability; Crossover; Ramipril
MeSH Terms: interventions — Ramipril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ramipril (Experimental): Ramipril 10 mg capsules of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Ramipril
- Altace (Active Comparator): Altace@ 10 mg capsules of Kings Pharmaceuticals, USA
  Interventions: Drug: Altace

INTERVENTIONS:
Drug: Ramipril — Ramipril 10 mg Capsules of Dr. Reddy's Laboratories Limited
  Other Names: Altace@10 mg Capsules
  Arms: Ramipril
Drug: Altace — Altace@ 10 mg capsules of Kings Pharmaceuticals, USA
  Arms: Altace

SUMMARY:
The purpose of this study is

* To characterize the pharmacokinetic profile of the Ramipril 10 mg capsules relative to that of ALTACE@ 10 mg capsules in healthy, adult, human, male subjects under fasting conditions and to assess the bioequivalence.
* To monitor the safety of the subjects.

DETAILED DESCRIPTION:
A Two-way open label crossover experimental evaluation of relative bioavailabilities of Ramipril 10 mg capsules of Dr.Reddy's Laboratories and ALTACE@ 10 mg capsules of King Pharmaceuticals in healthy adult human male subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males between 18 and 45 years of age (both inclusive) living in and around Ahmedabad city of western part of India.
2. Having a Body Mass Index (BMI) between 18.5 and 24.9 (both inclusive), calculated as weight in kg/height in m2
3. Not having any significant diseases or clinically significant abnormal findings during screening, medical history, physical examination, laboratory evaluations, ECG and X-ray recordings.
4. Able to comply with the study procedures, in the opinion of the investigator.
5. Able to give written consent for participation in the trial.

Exclusion Criteria:

1. Known hypersensitivity or idiosyncratic reaction to ramipril or any other related drugs.
2. Any disease or condition which might compromise the haemopoietic, renal, hepatic,endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological,gastrointestinal or any other body system.
3. Use of any medicine within 14 days prior to start of the study. In any such case subject selection will be at the discretion of the Principal Investigator/Medical expert
4. Any history or presence of asthma (including aspirin induced asthma)or nasal polyp.
5. A recent history of alcoholism < 2 years) or of moderate (180 mL/day) alcohol use, or consumption of alcohol within 48 hr prior to receiving IP.
6. Smokers, who smoke more than 10 cigarettes/day or inability to abstain from smoking during the study.
7. The presence of clinically significant abnormal laboratory values during screening.
8. Use of any recreational drugs or history of drug addiction or testing positive in pre-study drug scans.
9. History of psychiatric disorders.
10. A history of difficulty in donating blood.
11. Donation of blood (1 unit or 350 mL) within 90 days prior to receiving the first dose of IP.

    Note: In case, the blood loss was ≤ 200 mL, subject may be enrolled 60 days after the blood donation.
12. A positive hepatitis screen including hepatitis B surface antigen, Anti- HCV and Anti-HAV antibodies.
13. A positive test result for HIV antibody and/or syphilis.
14. The receipt of an investigational drug or product, or participation in a drug research study within a period of 90 days prior to the first dose of IP (Elimination half-life of the study drug should be taken into consideration for inclusion of the subject in the study).

    Note: If subject had participated in a study in which blood loss was ≤ 200 mL, subject can be dosed after completion of 60 days after the last sample of the previous study.
15. An unusual diet, for whatever reason (e.g. low-sodium), for four weeks prior to receiving the IP and throughout the subjects' participation in the study. In any such case subject selection will be at the discretion of the Principal Investigator/Medical expert.
16. Sitting blood pressure less than 110/70 mm Hg or pulse rate less than 60 or more than 100 beats per minute at screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2005-09; Primary Completion 2005-09 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Bioavailability based on Cmax and AUC parameters | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Mr. Charu Gautam, MD, DNB, Principal Investigator — Lambda Therapeutic Research Limited
Locations (1):
- Lambda Therapeutic Research Limited, Ahmedabad, Gujarat, India